CLINICAL TRIAL: NCT07369778
Title: Prospective Evaluation of Adler Laboratory's Massive Prosthetic Implants in Oncological and Non-oncological Situations
Acronym: IMPULSION
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0215
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Reconstruction of Massive Bone Loss (Oncologic and Non-oncologic)
Keywords: Megaprosthesis; pantheon; Massive bone loss
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Femur reconstruction Proximal (PFR)/Distal (DFR)/Total (TFR), Proximal Tibia (PTR), Custom implants: Massive prosthetic reconstruction using the Pantheon prosthesis from Adler Laboratories. The prostheses are:
  * Proximal Femur Recontruction (PFR)
  * Distal Femur Reconstruction (DFR)
  * Proximal Tibia Reconstruction (PTR)
  * Total Femur Reconstruction (TFR)
  * Custom implants

SUMMARY:
Massive prostheses are the standard treatment for extensive bone loss, whether caused by cancer or other factors (complex fractures, multiple revisions, infections).

The emergence of modular systems such as the Pantheon range provides rapid restoration of function and precise intraoperative adaptation to anatomical constraints and specific bone loss characteristics.

The Pantheon range also offers an innovative intramedullary ring system that promotes osseointegration and potentially long-term mechanical stability of implants.

However, few studies have evaluated its clinical efficacy. In this context, a prospective cohort study is warranted in order to obtain robust data on implant survival, patient quality of life and predictors of medium- and long-term complications.

DETAILED DESCRIPTION:
The IMPULSION study is an observational study. The primary objective is to evaluate prosthesis survival within 5 years post-operatively.

The secondary objectives are: to evaluate functional outcomes, quality of life, the occurrence of complications, and the osseointegration of the intramedullary ring.

Patients are included during the consultation to plan the surgery. Following surgery, the patient is followed up at 1 year, 2 years and 5 years post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 years or older at the time of inclusion
* Surgery scheduled at one of the participating centres with an Adler implant from the list below:

Implants from the Pantheon prosthesis:

Proximal Femur Recontruction (PFR) Distal Femur Reconstruction (DFR) Proximal Tibia Reconstruction (PTR) Total Femur Reconstruction (TFR) Hybrid connector implants Custom-made implants

* Follow-up scheduled at one of the participating centres for the duration of the study
* Patient who has been informed about the study and does not object to participating In the case of minor patients, the patient's parents will also be informed, and their non-objection will be sought.
* Patient affiliated with a Social Security scheme in France.

Exclusion Criteria:

* Patient or parent of a minor patient who objects to participation in the study and data collection.
* Patient deprived of liberty or under legal protection (guardianship or curatorship)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population concerns patients with massive bone loss, because of oncological or non-oncological issue. Patients have massive prosthetic reconstruction using the Pantheon prosthesis from Adler Laboratories. The prostheses are:
  * Proximal Femur Recontruction (PFR)
  * Distal Femur Reconstruction (DFR)
  * Proximal Tibia Reconstruction (PTR)
  * Total Femur Reconstruction (TFR)
  * Custom implants Minors aged 15 and over may be included in the study, with no maximum age limit. Patient who has been informed about the study and doesn't object to participating.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2036-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of prosthesis survival | 1 year, 2 years and 5 years post-operative
  The survival of the prosthesis is defined by the absence of revision surgery. This objective will be analysed in subgroups according to the type of implant used (PFR, DFR, PTR, TFR) or other implants (hybrid connector, custom-made).

SECONDARY OUTCOMES:
Evaluation of functional outcomes | 1 year after surgery (Y1), 2 years (Y2) and 5 years (Y5)
  MSTS score collected at inclusion, then post-operatively: 1 year after surgery (Y1), 2 years (Y2) and 5 years (Y5) As with the main objective, these objectives will be analysed in subgroups according to the type of implant used (PFR,DFR,PTR,TFR) or other implants (hybrid connector, custom-made).
Evaluation of quality of life | 1 year after surgery (Y1), 2 years (Y2) and 5 years (Y5)
  EQ-5D-5L auto-questionnaire at inclusion, then post-operatively: 1 year after surgery (Y1), 2 years (Y2) and 5 years (Y5) As with the main objective, these objectives will be analysed in subgroups according to the type of implant used (PFR,DFR,PTR,TFR) or other implants (hybrid connector, custom-made).
Evaluation of complications occurring within 5 years post-operatively | 1 year after surgery (Y1), 2 years (Y2) and 5 years (Y5)
  Complications coded according to the Henderson classification within 5 years post-operatively As with the main objective, these objectives will be analysed in subgroups according to the type of implant used (PFR,DFR,PTR,TFR) or other implants (hybrid connector, custom-made).
Evaluation of osseointegration of the intramedullary ring | 1 year after surgery (Y1), 2 years (Y2) and 5 years (Y5)
  Radiographic analysis 1 year after surgery (Y1), 2 years (Y2) and 5 years (Y5) (4 cortical images on front and profile views): osseointegration Yes/No/Don't know As with the main objective, these objectives will be analysed in subgroups according to the type of implant used (PFR,DFR,PTR,TFR) or other implants (hybrid connector, custom-made).

IPD SHARING:
Plan to Share IPD: No